CLINICAL TRIAL: NCT05788341
Title: The Israeli Study for Islet Autoantibodies Screening in Families of Type-1 Diabetes Patients
Status: Recruiting | Type: Observational
Sponsor: Rabin Medical Center (Other)
Collaborators: Provention Bio, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: RMC009523ctil
Record Dates: First submitted 2023-03-15; First posted 2023-03-28 (Actual); Last update posted 2024-03-27 (Actual); Status verified 2024-03

CONDITIONS: Type 1 Diabetes
Keywords: Stage 1 diabetes; stage 2 diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus

STUDY DESIGN:
Observational Model: Family Based | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
We aim at establishing a research program that will offer screening for the presence of Islet Autoantibodies (IA) in relatives of people with Type 1 Diabetes (T1D).

Relatives of people with diabetes, children, and adults from our clinic and all over Israel will be offered to participate in the study. The presence of IA will be evaluated using the Detection by Agglutination-PCR (ADAP) technology developed by Enable Biosciences, which is 1,000-10,000 times more analytically sensitive than currently used methods.. When positive in the screening, multiple antibodies will be confirmed by a second sample analyzed by the ADAP technology and by a radio binding assay (RBA). People positive for one or more antibodies (stage 1 or 2 T1D) will be referred to attend an educational program at our center. This program will include diabetes education emphasizing DKA prevention as well as stress assessment for the families involved and stress alleviating interventions. After the educational visit, people at risk of developing diabetes will be referred to further follow-up and evaluation under routine medical care at our center.

ELIGIBILITY:
Inclusion Criteria:

* First degree family member (sibling or parent) of a known T1D patient
* Age 2-45 years
* Signing an informed consent

Exclusion Criteria:

* Known diabetes of any kind (type 2, MODY)
* Have a previous history of being treated with insulin or oral diabetes medications.
* Currently be using systemic immunosuppressive agents (topical and inhaled agents are acceptable)

Ages: 2 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: First degree relatives of people with TID
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2023-05-30 (Actual); Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Positive Islet Autoantibodies | Screening visit

CONTACTS AND LOCATIONS:
Locations (1):
- Schneider Children Medical Center of Israel, Petah Tikva, Israel